CLINICAL TRIAL: NCT03238157
Title: Steroids for Early Treatment of Radiation Retinopathy
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Arun SINGH, Professor, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NDA 201923
Record Dates: First submitted 2017-07-31; First posted 2017-08-03 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Radiation Retinopathy
MeSH Terms: interventions — Fluocinolone Acetonide; Steroids

STUDY DESIGN:
Intervention Model Description: Randomized to either observation (2:1) (standard of care) or intravitreal Fluocinolone Acetonide (FA) implant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Observation (No Intervention): The study will only include those patients that are ascertained be at more than 50% risk for vision loss (20/200 or worse at 3 years) because of total radiation dose of >40 Gy to the center of the macula. These "at risk" patients included in the study will receive intravitreal triamcinolone (4 mg in 0.1 ml) injected at the time of plaque removal. If lack of IOP rise (30 mm Hg or more) at 3 months, then randomized to either observation (2:1) (standard of care).
- Intervention (Active Comparator): The study will only include those patients that are ascertained be at more than 50% risk for vision loss (20/200 or worse at 3 years) because of total radiation dose of >40 Gy to the center of the macula.1 These "at risk" patients included in the study will receive intravitreal triamcinolone (4 mg in 0.1 ml) injected at the time of plaque removal. If lack of IOP rise (30 mm Hg or more) at 3 months, then randomized to intravitreal Fluocinolone Acetonide (FA) implant.
  Interventions: Drug: Fluocinolone Acetonide (FA) implant

INTERVENTIONS:
Drug: Fluocinolone Acetonide (FA) implant — Fluocinolone Acetonide (FA) implant is designed to release FA at an initial rate of approximately 0.6 g/d, decreasing over the first month to a steady rate of 0.3 to 0.4 g/d with a duration of approximately 30 months.
  Other Names: Steroid
  Arms: Intervention

SUMMARY:
Radiation retinopathy is a known complication of ocular radiation therapy. To date there is no known effective treatment. In addition to their anti-vascular endothelial growth factor (VEGF) properties, corticosteroids decrease the retinal capillary permeability by increasing the activity/density of tight junctions and acute inflammatory effects of radiation in various tissues.

DETAILED DESCRIPTION:
The purpose of the project is threefold:

1. To study the natural history of radiation retinopathy using advanced imaging techniques. A combination of macular OCT to evaluate for edema, OCT angiography to evaluate for macular and peri-papillary ischemia and wide-field angiography for peripheral ischemia and leakage. Potential role of OCT angiography in radiation retinopathy will be evaluated by comparison to other eye (control) and FA.
2. Currently there is no consensus on effective management strategy for radiation retinopathy. Patients in the interventional will be prospectively followed to study efficacy of steroids for early treatment of radiation retinopathy while comparing the multimodal therapeutic approach in a randomized trial.
3. Patients in the observational arm will be prospectively followed while comparing the multimodal therapeutic approach in a randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Primary uveal melanoma
* Primary treatment with plaque brachytherapy
* Baseline visual acuity 20/200 or better
* Posterior tumor margin >1.50 mm from the center of the macula
* Posterior tumor margin > 1.50 mm from the closest disc margin
* Calculated total dose to center of the macula >40 Gy

Exclusion Criteria:

* Iris melanoma
* Opaque media
* less than 21 years of age
* Inability to give consent
* Positive pregnancy test

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Central subfield retinal thickness by OCT scan | 24 months
  Anatomic outcome

SECONDARY OUTCOMES:
Best corrected visual acuity | 24 months
  Functional outcome Best corrected Visual acuity and Visual field defect

OTHER OUTCOMES:
Need for standard of care intervention | 24 months
  standard of care intervention with laser photocoagulation and/ or anti VEGF agents

CONTACTS AND LOCATIONS:
Locations (1):
- Cole Eye Instiute, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided